CLINICAL TRIAL: NCT05941949
Title: An Examination Into the Effects of a Nutraceutical Supplement on Cognition, Stress, and Eye and Skin Health in Adults With Self-reported Cognitive Complaints: a Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Nutritional Supplement's Effects on Cognition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pharmanex (Industry)
Collaborators: Clinical Research Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PHX 1.2
Record Dates: First submitted 2023-05-26; First posted 2023-07-12 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Dietary Supplement; Cognition; Healthy
Keywords: Dietary Supplement; Cognition; Memory; Mental Stress; Wellbeing; Antioxidant; Astaxanthin; Grape Juice Extract
MeSH Terms: conditions — Stress, Psychological | interventions — astaxanthine; Olive Oil

STUDY DESIGN:
Intervention Model Description: Randomized, Prospective, Double Blind, Placebo-Controlled design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Softgels with similar appearance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Softgel containing: Astaxanthin, Grape Juice Extract, and All Natural Vitamin E
  Interventions: Dietary Supplement: Softgel Cognitive Formulation containing Astaxanthin, Grape Juice Extract and All Natural Vitamin E
- Placebo (Placebo Comparator): Softgel containing: Olive Oil and Sunflower Lecithin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Softgel Cognitive Formulation containing Astaxanthin, Grape Juice Extract and All Natural Vitamin E — 2 softgels per day
  Other Names: Astaxanthin, Grape Juice Extract, All Natural Vitamin E
  Arms: Active
Dietary Supplement: Placebo — 2 softgels per day
  Other Names: Olive oil
  Arms: Placebo

SUMMARY:
This is a prospective, placebo controlled study, examining the effects of dietary supplement's effects on cognition and confirming safety.

DETAILED DESCRIPTION:
The objective of this prospective, placebo controlled, double-blinded, parallel-group study is to examine the effects of dietary supplement containing grape juice extract, astaxanthin, and vitamin E over 12 week consumption on cognitive performance and self report results based on questionnaires. Furthermore, an evaluation of general well-being, mood, markers of oxidative stress, neurogenesis (BDNF), eye health, skin health, skin carotenoid concentrations, and safety measurements will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Health Individuals
* Residing in independent living accommodations
* Subjective report of memory or attention problems by answering 'yes' to the following questions: Do you have problems with your memory, attention, or concentration?
* Non-smoker
* Body Mass Index (BMI) between 18-35 kg/m2
* No plan to commence new treatments over the study period
* Understand, willing and able to comply with all study procedures
* Willing to provide a personally signed and dated informed consent form detailing all pertinent aspects of the study

Exclusion Criteria:

* Diagnosis of dementia based on the revised National Institute on Aging-Alzheimer's Association (NIA/AA) criteria
* A score below the 5th percentile for age, education, and gender on the Telephone Interview for Cognitive Status (TICS-M)
* Suffering from recently diagnosed or unmanaged medical conditions including but not limited to diabetes, hyper/hypotension, cardiovascular disease, gallbladder disease, autoimmune disease, endocrine disease, or cancer/malignancy
* Diagnosis of a psychiatric disease (other than mild-to moderate depression of anxiety) and/or neurological condition/disease (e.g. Parkinson's, Alzheimer's disease)
* History of paralysis, stroke or seizures or head injury (with loss of consciousness)
* Regular medication intake including but not limited to anticholinergics, acetylcholinesterase inhibiters, or steroid medications.
* Taking vitamins or herbal supplements that are reasonably expected to influence study measures
* In the last 6 month, commenced or changed the dose of nutritional and/or herbal supplements that may impact on treatment outcome
* Alcohol intake greater than 14 standard drinks per week
* Current or 12-month history of illicit drug abuse
* Pregnant women, women who are Brest feeding, or women who intend to fall pregnant
* Any significant surgeries over the last year
* Planned major lifestyle change in the next 3 months

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in working memory | Baseline and Week 12
  Determine change in working memory as measured by the Numeric Working Memory Test
Change in Working memory by Corsi Block tasks | Baseline and Week 12
  Determine if working memory change by doing Corsi blocks task
Change in verbal learning and memory | Baseline and Week 12
  Determine if verbal learning and memory change using total score on Rey Auditory Verbal Learning test trials 1 to 5
Change in episodic memory | Baseline and Week 12
  Determine change in episodic memory as measured by Rey Auditory Verbal Learning Test delayed recall and computerized location learning task

SECONDARY OUTCOMES:
Change in accuracy of attention | Baseline and Week 12
  Determine change inaccuracy of attention as measured by the choice reaction time and digit vigilance task (percent correct)
Change in the Everyday Memory | Baseline, Week 4, Week 8, Week 12
  Determine the change in the Everyday Memory Questionnaire total score
Change in the Perceived Stress score | Baseline, Week 4, Week 8, Week 12
  Determine the change in the Perceived Stress Questionnaire total score
Change in the World Health Organization score | Baseline, Week 4, Week 8, Week 12
  Determine the change in the World Health Organization-5 (WHO-5) score
Change in oxidative stress marker | Baseline and Week 12
  Determine change in plasma malondialdehyde
Change in plasma Tumor Necrosis Factor-alpha concentrations | Baseline and Week 12
  Determine change in plasma Tumor Necrosis Factor concentrations
Change in marker of inflammation in the plasma | Baseline and Week 12
  Determine the change in the plasma marker (interleukin-6-alpha concentrations
Change in plasma Brain-derived neurotropic factor concentrations | Baseline and Week 12
  Determine the change in plasma Brain-derived neurotropic factor concentrations
Change in Skin Carotenoid Score | Baseline and Week 12
  Determine the change in Skin Carotenoid Scores using Raman spectroscopy (BioPhotonic Scanner)

OTHER OUTCOMES:
Change in Ocular Surface Disease Index score | Baseline, Week 4, Week 8, Week 12
  Determine the change in Ocular Surface Disease Index score
Change in diastolic blood pressure measurement (safety measure) | Baseline and Week 12
  Determine change in diastolic blood pressure changes using sphygmomanometer
Change in systolic blood pressure measurement (safety measure) | Baseline and Week 12
  Determine change in systolic blood pressure measurement using sphygmomanometer

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Lopresti, MD, Principal Investigator — Clinical Research Australia
Locations (1):
- Clinical Research Australia, Duncraig, Western Austrailia, Australia

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data. Will only report summary data i.e. means by responses to specific variables.